CLINICAL TRIAL: NCT04172610
Title: The Prevalence of Influenza Related Invasive Aspergillosis in Swedish Intensive Care Units
Brief Title: Prevalence of Influenza RelAted Invasive Aspergillosis
Acronym: PIRAIA
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Krifors, Principal Investigator, Karolinska University Hospital
Other Study IDs: K 2019-9546
Record Dates: First submitted 2019-11-11; First posted 2019-11-21 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Invasive Pulmonary Aspergillosis; Influenza, Human
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter study with the aim to determine the prevalence of influenza-related invasive pulmonary aspergillosis in Swedish intensive care units and to assess the clinical impact of and risk factors for influenza-related invasive pulmonary aspergillosis

DETAILED DESCRIPTION:
This is a multicenter prospective observational study conducted at 12 intensive care units (ICU) in Sweden. All patients >18 years of age with a Polymerase Chain Reaction (PCR)-verified influenza A or B diagnosed up to 7 days before admission to the ICU or during ICU care, will be included in the study.

A new clinical routine has been implemented at the study centers: During the ICU stay screening with Beta-D-glucan and Galactomannan in blood/serum will be performed twice weekly and a respiratory sample will be retrieved for fungal culture and microscopy once weekly.

All results from collected samples will be available to the patient's attending physicians. Clinical and microbiological data will be collected, and the diagnosis of invasive aspergillosis will be made using predefined diagnostic criteria.

Objectives:

1. To determine the prevalence of influenza-related invasive pulmonary aspergillosis in Swedish intensive care units
2. To assess the clinical impact of and risk factors for influenza-related invasive pulmonary aspergillosis

ELIGIBILITY:
Inclusion Criteria:

* Confirmed influenza A or B diagnosed up to 7 days before ICU admission, or during ICU care
* Admitted to the ICU

Exclusion Criteria:

- Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients ≥18 years of age with confirmed influenza A or B diagnosed up to 7 days before ICU admission, or during ICU care, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of proven or probable invasive pulmonary aspergillosis | From date of enrollment up to 90 days after enrollment
  Enrolled patients will be categorized as proven or probable invasive pulmonary aspergillosis at discharge from the ICU.

SECONDARY OUTCOMES:
Sequential Organ Failure assessment Score (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Registered once daily. Range 0-24, a higher score indicates a higher mortality risk
Use of mechanical ventilation (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Yes/No. Registered once daily.
Use of non-invasive ventilation (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Yes/No. Registered once daily
Use of vasopressor (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not)pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Yes/No. Registered once daily.
Use of renal replacement therapy (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Yes/No. Registered once daily.
Acute Respiratory Distress Syndrome (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Registered once daily, using the Berlin-definition (mild 200 mm Hg < PaO2/FIO2 ≤ 300 mm Hg), moderate (100 mm Hg < PaO2/FIO2 ≤ 200 mm Hg), and severe (PaO2/FIO2 ≤ 100 mm Hg)
Days of ICU stay (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Median number of days
ICU mortality (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  Yes/No
90-day mortality after ICU admission (in patients diagnosed with proven/probable invasive pulmonary aspergillosis and those that were not) | from date of ICU admission to 90 days after ICU admission
  Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Anders Krifors, M.D., Principal Investigator — Karolinska Institutet; Markus Castegren, M.D. Ph.D., Study Director — Karolinska Institutet; Ola Blennow, M.D. Ph.D., Study Chair — Karolinska Institutet; Johan Petersson, M.D. A/Prof., Study Chair — Karolinska Institutet
Locations (12):
- Sweden (12):
  - ICU at Mälarsjukhuset, Eskilstuna
  - ICU at Helsingborgs lasarett, Helsingborg
  - ICU at Länssjukhuset Ryhov, Jönköping
  - ICU at Universitetssjukhuset, Linköping
  - ICU at Skånes universitetssjukhus, Lund
  - ICU at Skånes universitetssjukhus, Malmo
  - ICU at Universitetssjukhuset, Örebro
  - ICU at Danderyds sjukhus, Stockholm
  - ICU at Karolinska Universitetssjukhuset Huddinge, Stockholm
  - ICU at Karolinska Universitetssjukhuset Solna, Stockholm
  - ICU at Akademiska sjukhuset, Uppsala
  - ICU at Västmanlands sjukhus, Västerås

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Derived] Krifors A, Blennow O, Pahlman LI, Gille-Johnson P, Janols H, Lipcsey M, Kallman J, Tham J, Stjarne Aspelund A, Ljungquist O, Hammarskjold F, Hallgren A, De Geer L, Lemberg M, Petersson J, Castegren M. Influenza-associated invasive aspergillosis in patients admitted to the intensive care unit in Sweden: a prospective multicentre cohort study. Infect Dis (Lond). 2024 Feb;56(2):110-115. doi: 10.1080/23744235.2023.2273381. Epub 2023 Dec 18. PMID 37897800

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT04172610/Prot_SAP_000.pdf